CLINICAL TRIAL: NCT02488356
Title: Safety and Efficacy of Litramine IQP G-002AS for Weight Loss: A Randomised, Double-blind, Placebo-controlled, Parallel-group Study
Brief Title: Litramine for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InQpharm Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: INQP1200
Record Dates: First submitted 2015-06-30; First posted 2015-07-02 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Litramine (Experimental): Patented fibre complex from Opuntia ficus-indica (Litramine)
  Interventions: Dietary Supplement: Litramine
- Placebo (Placebo Comparator): Inert fillers that is manufactured to look and taste the same as verum
  Interventions: Dietary Supplement: Litramine

INTERVENTIONS:
Dietary Supplement: Litramine
  Other Names: IQP G-002AS

SUMMARY:
Safety and Efficacy of Litramine in weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects ≥18 and ≤ 60 years of age
* Body mass index (BMI) ≥ 25 and ≤35 kg/m2
* Judged by the Investigator to be in general good health on the basis of medical history
* Judged by the Investigator to be motivated to lose weight
* Accustomed to 3 main meals per day
* Consistent and stable body weight 3 months prior to study enrollment (±5%)
* Consistent regular physical activity
* Agree to stop all medications and supplements during the entire length of the study
* Commitment to adhere to diet and lifestyle recommended for the study
* Females of child bearing potential must agree to use appropriate birth control methods during the entire study period
* Stable concomitant medications
* Understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator

Exclusion Criteria:

* Presence of any active gastrointestinal disease

  * Malabsorption disorders
  * Pancreatitis
  * Stenosis in the GI tract
  * Bariatric surgery/Lapband and bypass surgery
  * Abdominal surgery within 6 months prior to the study
* Subjects whose weight increases 1.5 pounds from screening to the baseline visit
* History of eating disorders like bulimia, anorexia nervosa, binge-eating
* Renal conditions / disease, history of nephrolithiasis
* Cardiac diseases requiring drug therapy
* Other serious organ or systemic diseases such as diabetes mellitus, standard laundry list of cardiac diseases
* Osteoporosis or on medications for osteoporosis
* Known sensitivity to the ingredients of the study medication
* Vegetarian or Vegan
* Daily use of dietary supplement (2 week washout is allowed)
* Any medication that could influence gastrointestinal functions such as antibiotics, laxatives, opioids, anticholinergics, or anti-diarrheals (must have stopped at least 3 months before study start)
* Subjects who are pregnant or lactating
* Any medication or use of products for the treatment of obesity (e.g., Xenical, other fat binder, fat burner, satiety products etc.)
* Subjects who are currently on carbohydrate and protein diet, or low fat diet
* More than 3 hours of strenuous physical activity per week
* History of abuse of drugs, alcohol or medication
* Smoking cessation within the 6 months prior to this study
* Subjects unable to understand or follow the study protocol
* Participation in similar study or weight loss program within 6 months prior to this study
* Participation in other studies with in the last 4 weeks

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2012-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in body weight from baseline | 12 weeks